CLINICAL TRIAL: NCT00475657
Title: Phase II Study of Pemetrexed Plus Cisplatin in the Treatment of Patients With Extensive Small Cell Lung Cancer
Brief Title: Pemetrexed and Cisplatin as Treatment in Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11473; H3E-XM-S113
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Results first posted 2009-05-25 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: pemetrexed; Drug: cisplatin

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2, intravenous (IV), every 21 days x 6 cycles
  Other Names: LY231514; Alimta
Drug: cisplatin — 75 mg/m2, intravenous (IV), every 21 days x 6 cycles

SUMMARY:
The purpose of this study is to determine if cisplatin and pemetrexed are effective in the treatment of patients with Small Cell Lung Cancer, extended disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of Small Cell Lung Cancer (SCLC).
* Functional stage from 0 to 2 of the ECOG functional scale
* No previous systemic chemotherapy, immunotherapy or biologic therapy for SCLC.
* Previous bone marrow radiotherapy less than 25% is allowed.
* There must be at least one measurable lesion that complies with the solid tumor response evaluation criteria.
* Appropriate organic function.
* Life expectancy estimated at 12 weeks minimum.
* Females must be surgically sterile, postmenopausal or follow approved medical contraceptive methods during the treatment period and 6 months afterwards. Males must be surgically sterile or use a contraceptive method during the treatment period and during 6 months after treatment.
* The patient must be compliant and located close to the trial area for appropriate follow-up.
* The patient or his/her legal representative must sign an informed consent document.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Having received treatment for the last 30 days with a drug that has not obtained regulatory approval.
* Having participated in a previous pemetrexed trial.
* Mixed histologic diagnosis of SCLC and NSCLC.
* Concurrent illness.
* Having an active infection.
* Severe cardiac disease.
* Having received recently or concurrently a vaccine against yellow fever.
* Having suffered a previous malignant process other than SCLC.
* Central nervous system (CNS) metastases require concurrent corticoid therapy. Treated and stable CNS metastases are allowed.
* Clinically relevant fluid accumulation in the third space.
* Significant weight loss (greater than or equal to 10%) within 6 weeks prior to trial inclusion.
* Concurrent administration of any other anti-tumor treatment.
* Severe renal failure.
* Unable to discontinue administration of non-steroidal anti-inflammatory (NSAIDS) agents.
* Inability or unwillingness to take folic acid and vitamin B12 supplements.
* Inability to take corticoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Spain (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ferrol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lugo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ourense
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago de Compostela
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vigo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed + Cisplatin: Pemetrexed: 500 mg/m2, intravenous (IV), every 21 days x 6 cycles Cisplatin: 75 mg/m2, intravenous (IV), every 21 days x 6 cycles
Period: Overall Study
Arm/Group | Pemetrexed + Cisplatin
Started | 5
Completed | 1
Not Completed | 4
Not completed — Death | 1
Not completed — Sponsor's Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 66.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  Spain | 5
Race/Ethnicity [Number; unit: participants]
  Caucasian | 5
Height [Mean (Standard Deviation); unit: centimeters] | 163.9 (4.2)
Weight [Mean (Standard Deviation); unit: kilograms] | 76.0 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Trial terminated - results not analyzed
Time Frame: baseline to measured progressive disease
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: Trial terminated - results not analyzed
Time Frame: baseline to date of death from any cause
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression Free Survival
Description: Trial terminated - results not analyzed
Time Frame: baseline to measured progressive disease
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: Trial terminated - results not analyzed
Time Frame: time of response to progressive disease
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Stable Disease Rate
Description: Trial terminated - results not analyzed
Time Frame: baseline to measured progressive disease
Measure: Number; unit: participants
Arm/Group | Pemetrexed + Cisplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Pemetrexed + Cisplatin
Serious Adverse Events (participants affected / at risk) | 2
Other Adverse Events (participants affected / at risk) | 5
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Diarrhoea (Gastrointestinal disorders) | 1/5 (1)
Renal failure acute (Renal and urinary disorders) | 1/5 (1)
Pyrexia (General disorders) | 1/5 (1)
Dysphagia (Gastrointestinal disorders) | 1/5 (1)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed + Cisplatin
Anaemia (Blood and lymphatic system disorders) | 1/5 (1)
Asthenia (General disorders) | 1/5 (1)
Gamma-glutamyltransferase increased (Investigations) | 1/5 (1)
Blood creatine increased (Investigations) | 1/5 (1)
Leukopenia (Blood and lymphatic system disorders) | 1/5 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1/5 (1)
Nausea (Gastrointestinal disorders) | 1/5 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1/5 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1/5 (1)

LIMITATIONS AND CAVEATS:
On the advice of an independent monitoring board, this trial was stopped early due to lack of efficacy of the combination pemetrexed/carboplatin for small cell lung cancer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days